CLINICAL TRIAL: NCT06408155
Title: Improvement of Motor Tasks Performance: Effects of Verbal Encouragement and Music - Key Results From a Randomised Crossover Study With Electromyography
Brief Title: Improvement of Motor Tasks: Effects of Verbal Encouragement and Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Luca Puce, Principal Investigator, Universita degli Studi di Genova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DINOGMI-2024
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: motor recruitment; motivation; performance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Task with verbal encouragement (Experimental): Endurance isometric exercise performed with verbal encouragement
  Interventions: Other: Isometric Task
- Task 1 without motivational feedback (Active Comparator): Task without motivational feedback
  Interventions: Other: Isometric Task
- Task with music (Experimental): Endurance isometric exercise performed with music
  Interventions: Other: Isometric Task
- Task 2 without motivational feedback (Active Comparator): Task without motivational feedback
  Interventions: Other: Isometric Task

INTERVENTIONS:
Other: Isometric Task — The task demanded that participants maintain their arm bent at a 90° angle while holding a dumbbell, which weighed 80% of their one-repetition maximum (1RM), in a supine grip on the dominant side of their body for the longest time they could.

SUMMARY:
This study employed a randomized crossover design to assess the impacts of three different experimental conditions-standard environment, music, and verbal encouragement-on performance in an isometric endurance task, with comparisons made between untrained and trained individuals. Interventions were spaced seven days apart. Measurements included muscle activity and fatigue, assessed via surface electromyography, and the duration of the task.

The isometric endurance task required participants to maintain a 90° elbow flexion while holding a dumbbell in a supine grip, weighted to 80% of their one-repetition maximum, on the dominant side. During the task, participants were to keep their back and head against a vertical wall, stand with feet shoulder-width apart, and firmly on the ground. The dumbbell was held with the dominant arm, and the other arm was kept neutral by the side. It was crucial to avoid any rocking or movements that would ease maintaining the position. The test began when the bar was handed to the participant in the correct stance and concluded once the arm's angle deviated by more than five degrees from the start.

ELIGIBILITY:
Inclusion Criteria:

* Good general health,
* No medical conditions that could interfere with their ability to perform the test safely and effectively.
* To be considered exercised, participants had to have performed 150 minutes per week of vigorous intensity aerobic physical activity, in addition to muscle strengthening activities, for at least two days per week. Those who did not meet this standard were considered untrained.

Exclusion Criteria:

* History of surgery on the arm, shoulder or adjacent areas that could limit the ability to perform the test.
* Use of medication that affects muscle function or pain perception

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-13 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Duration of the task | Through task completion, an average of sixty seconds
  task duration expressed in seconds
Neuromuscular excitation of Biceps Brachii | Through task completion, an average of sixty seconds
  Amplitude of electromyography value (Root Mean Square in microvolt) measured for Biceps Brachii muscle
Neuromuscular excitation of Brachioradialis | Through task completion, an average of sixty seconds
  Amplitude of electromyography value (Root Mean Square in microvolt) measured for Brachioradialis muscle
Neuromuscular fatigue of Biceps Brachii | Through task completion, an average of sixty seconds
  Time-course evolution of the Median Frequency of the Power Density Spectrum (MF Hz) of the electromyography signal measured for biceps brachii muscle
Neuromuscular fatigue of Brachioradialis | Through task completion, an average of sixty seconds
  Time-course evolution of the Median Frequency of the Power Density Spectrum (MF Hz) of the electromyography signal measured for Brachioradialis muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Genova, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes